CLINICAL TRIAL: NCT00015236
Title: Modeling Impaired Judgement in Cocaine Abusers
Brief Title: Modeling Impaired Judgement in Cocaine Abusers - 6
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: New York MDRU (Other)
Masking: None | Purpose: Prevention
Other Study IDs: NIDA-5-0013-6; Y01-5-0013-6
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1998-06

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Amantadine

INTERVENTIONS:
Behavioral: Amantadine

SUMMARY:
The purpose of this study is for the modeling of impaired judgement in cocaine abusers.

DETAILED DESCRIPTION:
The objective of this study is to investigate recognition memory and appreciation of changing contingencies in relation to a response judgement.

ELIGIBILITY:
Inclusion Criteria:

(3 groups)Normal, healthy controls. Recent cocaine experience. Over 6 months since the last cocaine experience.

Exclusion Criteria:

Psychosis or mood disorder. History of seizure, head trauma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1997-03

CONTACTS AND LOCATIONS:
Overall Officials: John Rotrosen, M.D., Principal Investigator — New York MDRU
Locations (1):
- New York MDRU, New York, New York, United States

REFERENCES:
- [Background] NIDA Research Monograph Series 179, 1998 CPDD 98, 99.